CLINICAL TRIAL: NCT02821208
Title: Assessment and Prognostic Factors of Quality of Life in Patients With Psychogenic Nonepileptic Seizures
Brief Title: Quality of Life and Psychogenic Nonepileptic Seizures.
Acronym: PronoCNEP
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2014/04
Record Dates: First submitted 2016-06-22; First posted 2016-07-01 (Estimated); Last update posted 2022-05-13 (Actual); Status verified 2022-05

CONDITIONS: Psychogenic Nonepileptic Seizures (PNESs)
Keywords: Psychogenic nonepileptic seizure, quality of life
MeSH Terms: conditions — Psychogenic Nonepileptic Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- One cohorte : patient psychogenic nonepileptic seizures: The Psychogenic nonepileptic seizures (PNESs) are paroxysmal episodes type of abnormal movements, behavior modification or alteration of the contact-like seizures. These episodes are involuntary and underpinned by an unconscious psychological processes. In the International Classification of Disease-10 (ICD-10), they are classified as dissociative phenomena as conversing syndromes in the Manual of Diagnostic and Statistical Mental Disorders-IV (DSM-IV). The participants of the study only receive the usual care they would have if they were not included (no new/different intervention allocated in the study).

SUMMARY:
The goal of this study is to identify the prognostic factors of quality of life in patients with psychogenic non-epileptic seizures

DETAILED DESCRIPTION:
This is a monocentric prospective study. Our main objective is to identify prognostic factors associated with an improvement of quality of life on the QOLIE-31 and Short Form Health Survey "SF-36" at six months from the diagnostic.

We hypothesized that the absence of PNES during the last three-months before the six months follow-up visit is the best prognostic factor for an improvement of quality of life All adult (>15 years and 3 months) patients diagnosed with PNES will be prospectively included.

All patients will undergo standard of care and have consultation with neurologist and a psychiatrist trained for this type of disease, as it is usually made for these patients (no intervention allocated in the context of the research). . Announcement of diagnostic will be standardized and adapted to each patient. Clinical and demographic data will be collect as well as medical and psychiatric history. All patients will undergo prolonged electroencephalogram (EEG) under video monitoring allowing the diagnostic of PNES and ruling out epilepsy. Different neurologic and psychiatric scales will be collected (Quality of life in epilepsy - 31 quotes (QOLIE-31), Short Form Health Survey (SF-36), Montreal Cognitive Assessment (MoCA), Beck Depression Inventory (BDI2), Beck Anxiety index (BAI), Clinician administrated Post traumatic stress disorder scale (CAPS), Chilhood Trauma Questionnaire (CTQ), Epworth).

All patients will be oriented to psychiatric or psychological follow-up. Patients will undergo a one, three and six months follow-up and will be evaluated the number of seizure, their severity, and psychiatric or psychological follow-up will be evaluated. Patients will undergo scales (QOLI-31, SF-36, BDI2, BAI).

ELIGIBILITY:
Inclusion Criteria:

* Male or female adults (15 years and 3 months old)
* Psychogenic nonepileptic seizures (PNES) diagnosed as "probable" , "clinically established" or "documented" according to "Lafrance and al." criteria
* Having benefited a prolonged electroencephalogram recording under video control
* Patient Information and collection of non-opposition (patient or legal guardian)
* The patient or caregiver will be able to perform reliably the crisis diary and make the difference between PNES and epileptic seizure after investigator or co-investigator information.
* Affiliated to a social Insurance…

Exclusion Criteria:

* Patients for whom PNES have not been diagnosed
* Refused to participate
* The patient or his caregiver isn't able to perform reliably the crisis diary and don't make the difference between PNES and epileptic seizure after investigator or co-investigator information

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Every patient who come in hospital for diagnostic of Psychogenic nonepileptic seizures (PNES)
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2016-08-26 (Actual); Primary Completion 2020-06-12 (Actual); Study Completion 2020-06-12 (Actual)

PRIMARY OUTCOMES:
Improvement of the quality of life measured by the self-administered questionnaire QOLIE-31 (quality of life in epilepsy - QOLIE-31) | 6 months

SECONDARY OUTCOMES:
Average evolution in the quality of life measured by subscores of QOLIE -31 scale | 6 months
The average change in the quality of life, measured by the self-administered questionnaire SF -36 | 6 months
The proportion of patients with clinically significant improvement in quality of life subscores measured by the SF-36 | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Eric FRISON, Doctor, Study Chair — Unité de Soutien Méthodologique à la Recherche clinique et épidémiologique; University Hospital, Bordeaux
Locations (1):
- University Hospital of Bordeaux - Hospital Pellegrin, Bordeaux, France

IPD SHARING:
Plan to Share IPD: No